CLINICAL TRIAL: NCT03983135
Title: Results of Revisional Bariatric Surgery: A Single Center Experience
Brief Title: Revisional Bariatric Surgery Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Hakan Seyit, Medical Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BakırkoySadiKGeneralSurgery
Record Dates: First submitted 2019-05-26; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Bariatric Surgery; Revisional Bariatric Surgery; Obesity Associated Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients who undergo revisional bariatric surgery
  Interventions: Other: Laparoscopic mini gastric by-pass; Other: LaparoscopicRe-sleeve gastrectomy; Other: Laparoscopic Roux-en-Ygastric bypass

INTERVENTIONS:
Other: Laparoscopic mini gastric by-pass — Adhesions will separated along the left edge of the stomach and the left lobe of the liver. The remnant stomach will transected at the incisura angularis level with 60 mm Endo-GIA stapler(ATW 35, EthiconEndo-SurgeryInc., Cincinnati, OH, USA). Later ante-cholic distal of the Treitz ligament hadgastro-jejunal anastomosisof nearly 150 cm jejunal loop performed with 44 mm Endo-GIA stapler. Routinely, the omentum will be divided in two and omentopexy will be performed around the anastomosis. The stapler line will supported by absorbable stitches.
Other: LaparoscopicRe-sleeve gastrectomy — Adhesions will be separated with blunt and sharp dissections, then the remnant stomach will completely freed. Due to dilated antral pouch or fundus, the remnant stomach will resect as a tube stomach between the pillory and left crus with 60 mm Endo-GIA stapler accompanied by 36F bougie.
Other: Laparoscopic Roux-en-Ygastric bypass — all adhesions will separated then after the stomach pouch will formed by the linear stapler, 100 cm of jejunum will transected from the Treitz ligament. Side-to-side gastrojejunostomy will performed for the distal jejunum with the linear stapler. The anterior face of the anastomosis will manually sutured. Proximal jejunum end hadside-to-side jejuno-jejunostomy performed 150 cm distal of the gastrojejunostomy anastomosis with linear stapler on the posterior wall and manual suturing of the anterior wall.

SUMMARY:
The aim of this study is to assess the indications for revisional bariatric surgery and short-term revisional surgical outcomes such as weight loss, BMI variation, % excessive weight loss and % excessive BMI loss .Prospectively-collected patient data will retrospectively reviewed. Patient demographics, body mass index (BMI), primary and revision surgery types, indications of revision, outcomes of revisional surgery and follow-up data for comorbidities will investigated.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 65 years old,
* Patients who undergo revisional bariatric surgery due to renewed weight gain, stenosis or alkaline reflux after primary bariatric surgery

Exclusion Criteria:

* Eating disorders,
* Alcoholic
* Cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Weight loss (kilograms) | 3 years
  Amount of weight loss (kilograms) before (Day of surgery) and after (At three years) revisional bariatric surgery

SECONDARY OUTCOMES:
Resolution of comorbidities | 3 years
  The pharmacological treatment status of comorbidities related to obesity of type 2 diabetes (T2DM) and hypertension and gastroesophageal reflux will be observed with questions about "did it stop after surgery (improvement), did the dose or number of medications used reduce (resolution), or were there no changes?"comorbidities at the end of follow-up